CLINICAL TRIAL: NCT03037931
Title: A Randomized, Double-Blind, Placebo- Controlled Study to Investigate the Efficacy and Safety of Injectafer® (Ferric Carboxymaltose) as Treatment for Heart Failure With Iron Deficiency /and Sub-Study
Brief Title: Randomized Placebo-controlled Trial of FCM as Treatment for Heart Failure With Iron Deficiency / and Sub-Study
Acronym: HEART-FID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1VIT15043
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Iron-deficiency
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferric Carboxymaltose (Active Comparator): Ferric Carboxymaltose 2 doses intravenously of 15mg/kg to a maximum individual dose of 750mg 7 days apart and a maximum combined dose of 1500mg - repeated every 6 months as indicated by the results of iron indices.
  Interventions: Drug: Ferric Carboxymaltose
- Placebo (Placebo Comparator): Normal saline 15ml - 2 doses 7 days apart repeated every 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Carboxymaltose — Intravenous Iron
  Other Names: Injectafer, Ferinject
  Arms: Ferric Carboxymaltose
Drug: Placebo — Normal Saline Solution
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy and safety of iron therapy using intravenous (IV) ferric carboxymaltose (FCM), relative to placebo in the treatment of participants in heart failure with a reduced ejection fraction and with iron deficiency

DETAILED DESCRIPTION:
This is a double-blind, multicenter, prospective, randomized, placebo-controlled study to assess the effects of IV FCM compared to placebo on the 12-month rate of death, hospitalization for worsening heart failure, and the 6-month change in 6 minute walk test (6MWT) distance for patients in heart failure with iron deficiency.

After an initial screening period of up to 28 days, eligible participants will be stratified by region and randomized in a 1:1 ratio to FCM or placebo for treatment.

Study drug administration will occur on Day 0 and Day 7 (±2) as an undiluted slow IV push, with additional study visits planned at 3 month intervals, and additional dosing administered every 6 months as applicable. In a subset of sites, a sub-study will be conducted to characterize serum phosphate levels over time in participants with heart failure and iron deficiency after dosing with FCM. For all participants, hematology, ferritin, and transferrin saturation (TSAT), with appropriate safety evaluations, to determine additional treatment, will occur at 6 month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age) able to provide signed, written informed consent.
2. Stable heart failure (NYHA II-IV) on maximally-tolerated background therapy (as determined by the site Principle Investigator) for at least 2 weeks prior to randomization.
3. Able and willing to perform a six-minute walk test (6MWT) at the time of randomization.
4. Reduced left ventricular ejection fraction. Assessment must be performed at least 12 weeks after major cardiac surgical intervention including coronary artery bypass graft (CABG), valvular repair/replacement, or cardiac resynchronization therapy (CRT) device implantation.

   a. Left ventricular ejection fraction ≤ 40% obtained during the screening visit OR either of the following i. Historical value of ejection fraction ≤ 40% within 24 months of screening visit ii. Historical value of ejection fraction ≤ 30% within 36 months of screening visit
5. Hemoglobin >9.0 g/dL and < 13.5 g/dL (females) or <15.0 g/dL (males) within 28 days of randomization.
6. Serum ferritin <100 ng/mL or 100 to 300 ng/mL with TSAT <20%.Patients with screening ferritin <15 ng/mL must have documentation of an appropriate evaluation, as determined by the Principle Investigator, within 3 months of screening and prior to randomization.
7. Either documented hospitalization for heart failure within 12 months of enrollment or elavated N-terminal-pro-brain natriuretic peptide (NT-proBNP) within 90 days of randomization. a. For patients in normal sinus rhythm: N-terminal-pro-brain natriuretic peptide (NT- proBNP) > 600 pg/mL (or BNP >200 pg/mL) . b . For patients in atrial fibrillation: NT-proBNP >1000 pg/mL (or BNP >400 pg/mL) .

Exclusion Criteria:

1. Known hypersensitivity reaction to any component of FCM.
2. History of acquired iron overload, or the recent receipt (within 3 months) of erythropoietin stimulating agent, IV iron therapy, or blood transfusion.
3. Acute myocardial infarction, acute coronary syndrome, transient ischemic attack, or stroke within 30 days of enrollment.
4. Uncorrected severe aortic stenosis, severe valvular regurgitation (except mitral regurgitation due to left ventricular dilatation without planned intervention), or left ventricular outflow obstruction requiring intervention.
5. Current atrial fibrillation or atrial flutter with a mean ventricular response rate >100 per minute (at rest).
6. Current or planned mechanical circulatory support or heart transplantation.
7. Hemodialysis or peritoneal dialysis (current or planned within the next 6 months).
8. Documented liver disease, or active hepatitis (i.e. alanine transaminase or aspartate transaminase >3 times the upper limit of normal range).
9. Current or recent (within 3 years) malignancy with exception of basal cell carcinoma or squamous cell carcinoma of the skin, or cervical intraepithelial neoplasia.
10. Active gastrointestinal bleeding.
11. Female participant of child-bearing potential who is pregnant, lactating, or not willing to use adequate contraceptive precautions during the study and for up to 5 days after the last scheduled dose of study medication.
12. Inability to return for follow up visits within the necessary windows
13. Concurrently in a study with investigational product.
14. No participants with Current Coronavirus Disease-19 (COVID-19) Infection into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3065 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian F Hernandez, MD, Study Chair — Duke Clinical Research Institute
Locations (345):
- United States (188):
  - Advanced Cardiovascular LLC, Alexander City, Alabama
  - Advanced Cardiovascular, LLC, Auburn, Alabama
  - IMC/Diagnostic & Medical Clinic, Mobile, Alabama
  - University of South Alabama, Mobile, Alabama
  - Alaska Heart & Vascular Institute, Anchorage, Alaska
  - Verde Valley Medical Center, Cottonwood, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - Carondelet Heart and Vascular Institute - Cardiology East, Tucson, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Harbor-UCLA Medical Center, Carson, California
  - Valley Clinical Trials, Inc., Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - California Heart Specialists, Huntington Beach, California
  - First Valley Medical Group, Lancaster, California
  - Healthcare Partners Affiliation Medical Group, Long Beach, California
  - Axis Clinical Trials, Los Angeles, California
  - St. Joseph Heritage-Healthcare, Mission Viejo, California
  - Radin Cardiovascular Medical Group, Inc., Newport Beach, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Pasadena Clinical Research, Pasadena, California
  - Eugene Soroka, MD Inc., Port Hueneme, California
  - VA San Diego Health Care System, San Diego, California
  - Interventional Cardiology Medical Group, West Hills, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Christiana Care, Newark, Delaware
  - Alfieri Cardiology, Wilmington, Delaware
  - Cardiology Associates of South Florida, Boynton Beach, Florida
  - Cardiovascular & Vein Center of Florida, Bradenton, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - St. Vincent's Healthcare - Riverside, Jacksonville, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - St. Vincent's Healthcare - Southside Recruiting, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - ProLive Medical Research, Miami, Florida
  - Cordova Research Institute, LLC, Miami, Florida
  - Med-Care Research, Miami, Florida
  - ITB Research, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Empire Clinical Research, LLC, Miami Lakes, Florida
  - Florida Hospital Transplant Institute, Orlando, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Springfield Medical Center, Panama City, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - South Florida Research Solutions, LLC, Pembroke Pines, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Piedmont Heart Institute - Athens, Athens, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - University Cardiology Associates, LLC, Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - Piedmont Heart Institute Fayetteville, Fayetteville, Georgia
  - Georgia Arrhythmia Consultants and Research Institute, Macon, Georgia
  - Mercer University, Macon, Georgia
  - Atlanta Vanguard Research Institute, Smyrna, Georgia
  - Saint Luke's Boise Medical Center, Boise, Idaho
  - Mount Sinai Hospital Medical Center - Department of Cardiology, Chicago, Illinois
  - Medicoricium, LLC, Fairview Heights, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Franciscan Physician Network - Indiana Heart Physicians, Indianapolis, Indiana
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Indiana University Health Ball Memorial Hospital, Inc., Muncie, Indiana
  - Reid Physician Associates / Reid Health, Richmond, Indiana
  - Beacon Medical Group Advanced Cardiovascular Specialists, South Bend, Indiana
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Tulane Heart & Vascular Institute, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Maine Medical Partners Maine Health Cardiology, Scarborough, Maine
  - Anne Arundel Health System Research Institute, Annapolis, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NECCR Prima Care Research, LLC, Fall River, Massachusetts
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Western Michigan University Homer Stryker M.D. School of Medicine, Kalamazoo, Michigan
  - Michigan CardioVascular Institute at Covenant Medical Center, Saginaw, Michigan
  - Allina Health System, dba Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - North Kansas City Hospital, North Kansas City, Missouri
  - St. Louis Heart & Vascular, PC, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - CHI Health Research Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Red Rock Clinical Research, LLC, Las Vegas, Nevada
  - Monmouth Cardiology Associates, LLC, Eatontown, New Jersey
  - Englewood Health, Englewood, New Jersey
  - Advanced Heart & Vascular Institute of Hunterdon, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Trinity Medical WNY, PC, Cheektowaga, New York
  - Mount Sinai Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Richmond University Medical Center, Staten Island, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Circuit Clinical, West Seneca, New York
  - Northtowns Cardiology, PLLC, Williamsville, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Duke University Heart Failure Research, Durham, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Wake Forest University Health Sciences, High Point, North Carolina
  - Duke Cardiology of Lumberton, Lumberton, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Crossroads Clinical Research, Inc., Mooresville, North Carolina
  - Pinehurst Medical Clinic, Inc., Pinehurst, North Carolina
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - WakeMed Health and Hospitals, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Trinity Health Center - Medical Arts, Minot, North Dakota
  - Aultman Cardiology Clinical Trials, Canton, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - North Ohio Heart Center, Elyria, Ohio
  - North Ohio Heart Center, Sandusky, Ohio
  - Heart House Research Foundation, Springfield, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Health Holy Spirit Medical Center Geisinger - Cardiology, Camp Hill, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - V.A. Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Prisma Health, Columbia, South Carolina
  - Self Regional Hospital Research Center, Greenwood, South Carolina
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Black Hills Cardiovascular Research, a department of Rapid City Regional Hospital, Inc., Rapid City, South Dakota
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - Parkway Cardiology Associates, PC, Oak Ridge, Tennessee
  - Amarillo Hearth Clinical Research Institute, Inc., Amarillo, Texas
  - PharmaTex Research, Amarillo, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Texas Health Research & Education Institute, Fort Worth, Texas
  - Texas Heart Institute, Houston, Texas
  - Houston Heart & Vascular Associates, Kingwood, Texas
  - Caprock Cardiac Center Research Institute, Inc., Lubbock, Texas
  - Angelina Medical Research, LLC, Lufkin, Texas
  - North Dallas Research Associates, McKinney, Texas
  - North Texas Research Associates, McKinney, Texas
  - South Texas Cardiovascular Consultants, PLLC, San Antonio, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - PharmaTex Research, Tyler, Texas
  - The University of Texas Health Center at Tyler, Tyler, Texas
  - Wichita Falls Heart Clinic, Wichita Falls, Texas
  - Advanced Clinical Research/Intermountain Heart Center PC, West Jordan, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Riverside Cardiology Specialists, Newport News, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Hunter Holmes McGuire V.A. Medical Center - Cardiology Div. (111J), Richmond, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Swedish Heart & Vascular-Advanced Cardiac Support Program, Seattle, Washington
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington
  - CHI Franciscan Research Center, Tacoma, Washington
  - Walla Walla Clinic, Walla Walla, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth Care Inc / Waukesha Memorial Hospital, Waukesha, Wisconsin
- Australia (16):
  - SWSLHD-Liverpool Hospital, Liverpool, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Cairns Hospital, Cairns, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Core Research Group, Milton, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - SA Heart, Ashford, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Heart Lung Clinic, Darlinghurst, Sydney
  - Royal Hobart Hospital, Hobart, Tasmania
  - Royal Adelaide Hospital, Adelaide
  - Macquarie University - Clinical Trials Unit, Macquarie Park
  - John Hunter Hospital, New Lambton Heights
  - Epworth HealthCare Clinical Trials, Richmond
- Bulgaria (14):
  - MHAT Puls, Blagoevgrad
  - Multiprofile Hospital for Active Treatment: Department of cardiology, Gabrovo
  - MHAT Haskovo AD, Haskovo
  - Diagnostic - Consultative Center 1 - Lom - EOOD Office of Cardiology, Lom
  - Medical Center Medconsult Pleven OOD, Pleven
  - МC Hipokrena, Sevlievo
  - Diagnostic - Consultative Center XXII - Sofia EOOD, Office of Cardiology, Sofia
  - Second Medical Center-Sofia, EEOD - Department of Cardiology, Sofia
  - Second Multiprofile Hospital for Active Treatment, Sofia
  - 5th City Hospital, Sofia
  - National Multiprofile Transport Hospital Cardiology Clinic, Sofia
  - Medical Center Hera EOOD - Office of Cardiology, Sofia
  - Multiprofile Regional Hospital for Active Treatment, Veliko Tarnovo
  - Medical Center Velingrad 2017" EOOD, Office of Cardiology, Velingrad
- Canada (25):
  - University of Calbary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - South Edmonton Cardiology Consultants, Edmonton, Alberta
  - Royal Alexandria Hospital, Edmonton, Alberta
  - Fraser Clinical Trials, New Westminster, British Columbia
  - SMH Cardiology Clinical Trials, Surrey, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - G.A. Research Associates, Ltd., Moncton, New Brunswick
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Manna Research Inc., Burlington South, Burlington, Ontario
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - Vizel Cardiac Research, Cambridge, Ontario
  - London Health Sciences Center (LHSC), London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sinai Health System - Mount Sinai Hospital, Toronto, Ontario
  - Clinique de Cardiologie de Lévis, Lévis, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec - Université Laval, Québec, Quebec
  - CISSS de Chaudière-Appalaches (CISSS-CA), site Hôpital St-Georges, Saint-Georges, Quebec
  - Recherche Medical St-Jerome Inc., Saint-Jérôme, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux de la Mauricie-et-du-centre-du-Quebec, Trois-Rivières, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (7):
  - Interni kardiologicka klinika FN Brno, Brno
  - Kardiologicka ambulance, Chlumec nad Cidlinou
  - Centrum preventivní kardiologie, Karlovo nám. 32,, Prague
  - Centrum preventivní kardiologie, Prague
  - General University Hospital in Prague, Prague
  - General University Hospital, Prague
  - IKEM-Klinika kardiologie, Prague
- Georgia (10):
  - JSC Evex Hospitals,Georgia, Batumi
  - Clinic-LJ, Kutaisi
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - Ltd Israel-Georgian Medical Research Clinic "Helsicore", Tbilisi
  - Ltd Pineo Medical Ecosistem, Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center, Tbilisi
  - Bokhua Memorial Cardiovascular Center, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
  - Ltd TIM- Tbilisi Institute of Medicine, Tbilisi
  - Georgian-Dutch Hospital, Tbilisi
- Hungary (10):
  - Semmelweis Egyetem Városmajori Szív és- Érgyógyászati Klinika Szent Rókus Klinikai Tömb, Kardiológiai, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászati Klinika, Budapest
  - Debreceni Egyetem Klinikai Központ Kardiológiai Osztály, Debrecen
  - Clinexpert Gyöngyös Kft, Gyöngyös
  - Zsigmondy Vilmos Harkányi Gyógyfürdȍ Kórház, Harkány
  - Bács-Kiskun Megyei Kórház Kardiológiai Osztály, Kecskemét
  - Andrea Hornyik, MD, Miskolc
  - Pécsi Tudomány Egyetem Klinikai Központ, I. sz. Belgyógyászati Klinika,, Pécs
  - Jász-Nagykun-Szolnok Megyei Hetény i Géza Kórház Kardiológiai Osztály, Szolnok
  - Belvárosi Egészségház Kft, Zalaegerszeg
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Liepajas Regional Hospital, Liepāja
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East University hospital clinic Gailezers, Riga
- Lithuania (3):
  - The Hospital of Lithuanian, Kaunas
  - Klaipeda Seaman's Hospital, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- New Zealand (14):
  - Wellington Hospital, Newton, Wellington Region
  - Totara Clinical Research, Health New Lynn, Auckland
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Heart Institute, Christchurch
  - Dunedin Hospital, Dunedin
  - Hauora Tairāwhiti Department of Cardiology, Gisborne
  - Hawke's Bay Hospital, Hastings
  - Hutt Hospital, Lower Hutt
  - Nelson Hospital, Nelson
  - Taranaki Base Hospital, New Plymouth
  - Rotorua Hospital, Rotorua
  - Clinical Horizons NEW ZEALAND LTD, Tauranga
- Poland (16):
  - Oddział Kardiologii WSzS nr 4, Bytom
  - Biokinetica S.A. Przychodnia Józefów, Józefów
  - Centrum Medyczne Linden, Krakow
  - Marcin Ogórek, MD, PhD, Lodz
  - 1 Wojskowy Szpital Klininiczny w Lublinie, Lublin
  - Ko-Med Centra Kliniczne, Lublin
  - Szpital Swietej Anny w Miechowie, Miechów
  - Szpital Świętej Anny w Miechowie, Miechów
  - Nowodworskie Centrum Medyczne. Ambulatoryjna Opieka Specjalistyczna, Nowy Dwór Mazowiecki
  - Zespol Opieki Zdrowotnej, Oława
  - Wojewódzki Szpital Zespolony im. L. Rydygiera,Oddzialu Kardiologii i lntensywnej Terapii Kardiologicznej, Torun
  - Uniwersyteckie Centrum Kliniczne, Warsaw
  - Centrum Medyczne K2J2, Wołomin
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw
  - 4th Military Hospital, Wroclaw
  - Proximum Centrum Usług Medycznych NZOZ, Wroclaw
- Russia (14):
  - Municipal Autonomous Healthcare Institution "City Clinical Hospital #6, Chelyabinsk
  - Municipal Autonomous Healthcare Institution, Chelyabinsk
  - Federal State Budgetary Scientific Institution Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo
  - State Budgetary Healthcare Institution of Moscow city "Moscow, Moscow
  - Private Medical Institution "Euromedservice, Pushkin
  - State Budgetary Institution of Ryazan Region, Ryazan
  - JSC Polyclinic Complex, Saint Petersburg
  - Saint Petersburg Research Institute of Emergency Medicine n.a. I.I. Dzhanelidze, Saint Petersburg
  - Saint Petersburg Research Institute of Emergency Medicine, Saint Petersburg
  - LLC X7 Clinical Research, Saint Petersburg
  - Saint-Petersburg State Budgetary Institution of Healthcare "Saint Martyr Elizabeth city hospital", Saint Petersburg
  - LLC "Scientific Research Center Eco-Safety", Saint Petersburg
  - State Healthcare Institution, Saratov
  - Federal State Budget Educational Institution of Higher Education Saratov State Medical University of the Ministry of Health of Russia, Saratov
- Ukraine (24):
  - Municipal non-profit enterprise "Ivano-Frankivsk Regional Clinical Cardiological Center", Ivano-Frankivsk
  - Military and Medical Clinical Center of the Northern Region (Military Unit A-3306) Cardiology Department, Kharkiv
  - Scientific Medical Complex "University Clinic" of Kharkiv, Kharkiv
  - MNCE "City Hospital № 8" of Kharkiv City Council, Cardiology Department №2, Kharkiv
  - Communal Institution "Kryvyi Rih City Hospital №9" of Kryvyi Rih City Council, Kryvyi Rih
  - Municipal Non-Profit Enterprise "Consultative and Diagnostic centre" of Pechersk District of Kiyv, Kyiv
  - "Oleksandrivska Clinical Hospital of Kyiv" of executive authority Kyiv City, Kyiv
  - Communal nonprofit enterprise "Oleksandrivska Clinical Hospital of Kyiv, Kyiv
  - Communal non-profit enterprise Kyiv City Clinical Hospital №1, Kyiv
  - Kyiv City Clinical Hospital of Emergency Aid,, Kyiv
  - Kyiv City Clinical Hospital of Emergency Aid, Kyiv
  - Kyiv Clinic Railway Hospital №2 of the "Health Care Center" Brach at the PJSC "Ukrainian Railway", Kyiv
  - National Scientific Center Institute of Cardiology of M.D, Kyiv
  - State Institution "National Scientific Center "Institute of Cardiology, Kyiv
  - Medical Centre of LLC "Medical Centre "CONSILIUM MEDICAL", Kyiv
  - Medical Centre of LLC, Kyiv
  - MNPE "Lviv City Clinical Hospital No.5", Lviv
  - Communal Noncommercial Enterprise of Lviv Regional Council "Lviv Regional Clinical, Lviv
  - Vinnytsia Regional Clinical Hospital of Veterans of War, Vinnytsia
  - "Vinnytsia Regional Clinical Treatment Diagnostic Center of Cardiovascular Pathology", Vinnytsia
  - Communal Non-Profit Enterprise "City, Zaporizhzhia
  - Educational and Research Medical Center "University Clinic" at Zaporizhzhia State Medical University of the Ministry of Health of Ukraine,, Zaporizhzhia
  - Сommunal Institution "Zaporizhzhia Regional Clinical Hospital" of Zaporizhzhia Regional Council,, Zaporizhzhia
  - Communal Enterprise "Hospital №1" of Zhytomyr City Council, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis GD, Giczewska A, Mentz RJ, Butler J, Ezekowitz JA, De Pasquale C, O'Meara E, Troughton RW, Ponikowski P, Wong YW, Ikoma T, Malhotra R, Blackman N, Rockhold FW, Hernandez AF; HEART-FID Trial Investigators. Functional and Prognostic Implications of Different Iron Deficiency Definitions in Heart Failure: Insights From HEART-FID. JACC Heart Fail. 2025 Dec;13(12):102661. doi: 10.1016/j.jchf.2025.102661. Epub 2025 Oct 25. PMID 41137844
- [Derived] Harrington J, Mentz RJ, Rockhold FW, Garg J, Butler J, De Pasquale CG, Ezekowitz JA, Lewis GD, O'Meara E, Ponikowski P, Troughton RW, Wong YW, Adamczyk R, Storie T, Blackman N, Hernandez AF. Hierarchical End Points in Prior Heart Failure Trials and the HEART-FID Trial. Circ Heart Fail. 2024 Feb;17(2):e010676. doi: 10.1161/CIRCHEARTFAILURE.123.010676. Epub 2024 Jan 22. PMID 38250799
- [Derived] Mentz RJ, Garg J, Rockhold FW, Butler J, De Pasquale CG, Ezekowitz JA, Lewis GD, O'Meara E, Ponikowski P, Troughton RW, Wong YW, She L, Harrington J, Adamczyk R, Blackman N, Hernandez AF; HEART-FID Investigators. Ferric Carboxymaltose in Heart Failure with Iron Deficiency. N Engl J Med. 2023 Sep 14;389(11):975-986. doi: 10.1056/NEJMoa2304968. Epub 2023 Aug 26. PMID 37632463
- [Derived] Harrington J, Mentz RJ, Rockhold FW, Garg J, Butler J, De Pasquale CG, Ezekowitz JA, Lewis GD, O'Meara E, Ponikowski P, Troughton RW, Wong YW, Adamczyk R, Blackman N, Hernandez AF. Baseline characteristics of patients in the randomized study to investigate the efficacy and safety of ferric carboxymaltose as treatment for heart failure with iron deficiency: HEART-FID trial. Am Heart J. 2023 Dec;266:25-31. doi: 10.1016/j.ahj.2023.08.005. Epub 2023 Aug 19. PMID 37598795
- [Derived] Mentz RJ, Ambrosy AP, Ezekowitz JA, Lewis GD, Butler J, Wong YW, De Pasquale CG, Troughton RW, O'Meara E, Rockhold FW, Garg J, Samsky MD, Leloudis D, Dugan M, Mundy LM, Hernandez AF; HEART-FID Trial Investigators. Randomized Placebo-Controlled Trial of Ferric Carboxymaltose in Heart Failure With Iron Deficiency: Rationale and Design. Circ Heart Fail. 2021 May;14(5):e008100. doi: 10.1161/CIRCHEARTFAILURE.120.008100. Epub 2021 May 18. PMID 34003690

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferric Carboxymaltose | Placebo
Started | 1532 | 1533
Completed | 1123 | 1121
Not Completed | 409 | 412
Not completed — Death | 354 | 367
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 48 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose | Placebo | Total
Number analyzed (Participants) | 1532 | 1533 | 3065
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 508 | 525 | 1033
  >=65 years | 1024 | 1008 | 2032
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.57 (10.94) | 68.57 (11.20) | 68.57 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 506 | 531 | 1037
  Male | 1026 | 1002 | 2028
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85 | 100 | 185
  Not Hispanic or Latino | 1440 | 1424 | 2864
  Unknown or Not Reported | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 5 | 11
  Asian | 19 | 21 | 40
  Native Hawaiian or Other Pacific Islander | 6 | 5 | 11
  Black or African American | 162 | 160 | 322
  White | 1324 | 1325 | 2649
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  Hungary | 11 | 17 | 28
  United States | 612 | 601 | 1213
  Czechia | 14 | 19 | 33
  Ukraine | 243 | 217 | 460
  Russia | 58 | 65 | 123
  New Zealand | 46 | 54 | 100
  Canada | 109 | 120 | 229
  Latvia | 1 | 3 | 4
  Poland | 83 | 87 | 170
  Georgia | 88 | 92 | 180
  Australia | 59 | 51 | 110
  Bulgaria | 195 | 197 | 392
  Lithuania | 13 | 9 | 22
  Estonia | 0 | 1 | 1
Intent-to-treat Analysis Population [Count of Participants; unit: Participants] | 1123 | 1121 | 2244

OUTCOME MEASURES:

1. Primary Outcome: Number of Deaths
Description: The number of participants who died out of the total treated group.
Time Frame: 1 year
Population: Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 1532 | 1533
Participants | 131 | 158

2. Primary Outcome: Number of Hospitalizations for Heart Failure
Description: The number of participants who were hospitalized for heart failure out of the total treated group.
Time Frame: 1 year
Population: Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 1532 | 1533
Participants | 297 | 332

3. Primary Outcome: Change in 6MWT (Six Minute Walk Test) Distance
Description: The change in meters walked at baseline compared to 6 months later.
Time Frame: 6 months
Population: Number of participants within the ITT population which contributed to the 6MWT data
Measure: Mean (Standard Deviation); unit: unit of measure in meters
Arm/Group | Ferric Carboxymaltose | Placebo
Number analyzed (Participants) | 1285 | 1295
unit of measure in meters | 8.179 (59.963) | 3.979 (58.896)

ADVERSE EVENTS:
Time Frame: 67.5 months
Description: Adverse Events (AEs) specified in the protocol were collected for duration of study (67.5 max months duration). After early/permanent discontinuation AEs were reported for 30 days after study drug.
  Death for any cause was part of the composite primary endpoint. All mortality (Cardiovascular and all other causes) were collected for the duration of the study (67.5 max months duration). The mortality data is used in various secondary endpoint evaluations.
Arm/Group | Ferric Carboxymaltose | Placebo
All-Cause Mortality (participants affected / at risk) | 354/1532 | 367/1533
Serious Adverse Events (participants affected / at risk) | 413/1532 | 401/1533
Other Adverse Events (participants affected / at risk) | 424/1532 | 412/1533
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Carboxymaltose (N=1532) | Placebo (N=1533)
Pneumonia (Infections and infestations) | 57 (64) | 35 (37)
COVID-19 (Infections and infestations) | 39 (39) | 37 (39)
Sepsis (Infections and infestations) | 21 (22) | 13 (14)
Cellulitis (Infections and infestations) | 12 (12) | 21 (27)
COVID-19 pneumonia (Infections and infestations) | 11 (11) | 17 (17)
Urinary Tract Infection (Infections and infestations) | 17 (20) | 9 (11)
Osteomyelitis (Infections and infestations) | 7 (8) | 3 (3)
Influenza (Infections and infestations) | 5 (5) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4)
Septic shock (Infections and infestations) | 6 (7) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2) | 4 (4)
Localised infection (Infections and infestations) | 3 (4) | 2 (2)
Pyelonephritis (Infections and infestations) | 3 (3) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 2 (2)
Diabetic foot infection (Infections and infestations) | 1 (2) | 3 (5)
Urosepsis (Infections and infestations) | 4 (4) | 0 (0)
Appendicitis (Infections and infestations) | 1 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (3)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Implant site infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection staphylococcal (Infections and infestations) | 1 (2) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Candida pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Large intesting infection (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fascities (Infections and infestations) | 1 (1) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitiis acute (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (2)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sialoadentitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (14) | 15 (17)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 8 (10)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 6 (6)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 8 (8) | 11 (12)
Angina pectoris (Cardiac disorders) | 3 (3) | 8 (8)
Atrial Fibrillation (Cardiac disorders) | 5 (5) | 6 (6)
Ventricular tachycardia (Cardiac disorders) | 7 (7) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 6 (7) | 3 (4)
Angina unstable (Cardiac disorders) | 0 (0) | 6 (6)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 3 (3)
Cardogenic shock (Cardiac disorders) | 2 (2) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 3 (3)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 3 (3)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular dyssynchrony (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 9 (10)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (5) | 10 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (8) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Gout (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sycope (Nervous system disorders) | 11 (11) | 10 (10)
Metabolic encephalopathy (Nervous system disorders) | 2 (3) | 6 (6)
Presynope (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Encephalopathy (Nervous system disorders) | 3 (3) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 4 (4)
Seizure (Nervous system disorders) | 2 (2) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Radiculopathy (Nervous system disorders) | 2 (2) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 2 (2) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 2 (3)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial spasm (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Vascular demetia (Nervous system disorders) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 17 (17) | 14 (17)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 4 (4)
Hypertensive crisis (Vascular disorders) | 3 (3) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Giant cell arteritis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (2)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 10 (13) | 10 (11)
Asthenia (General disorders) | 4 (5) | 4 (4)
Chest pain (General disorders) | 3 (3) | 5 (6)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Medical device site haematoma (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pacemaker generated arrhythmia (General disorders) | 0 (0) | 1 (1)
Physical deconditioning (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (3)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocyctic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 15 (15)
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5) | 3 (4)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 1 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 3 (3) | 4 (4)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 2 (2)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (2)
Cardiac pacemaker evaluation (Investigations) | 0 (0) | 1 (1)
Cardiac stress abnormal (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
International normalised ration increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Transplant evaluation (Investigations) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 4 (4) | 3 (5)
Delirium (Psychiatric disorders) | 3 (4) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium febrile (Psychiatric disorders) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 2 (2)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Throidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Eye disorders (Surgical and medical procedures) | 2 (2) | 4 (4)
Cataract (Surgical and medical procedures) | 1 (1) | 1 (1)
Diplopia (Surgical and medical procedures) | 0 (0) | 1 (1)
Neovascular age-related macular degeneration (Surgical and medical procedures) | 0 (0) | 1 (1)
Retinal artery occlusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Heart transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo positional (Immune system disorders) | 0 (0) | 1 (1)
Device electrical finding (Product Issues) | 1 (1) | 0 (0)
Device electrial impedance issue (Product Issues) | 1 (1) | 0 (0)
Device power source issue (Product Issues) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 46 (60) | 40 (49)
Chronic kidney disease (Renal and urinary disorders) | 8 (8) | 5 (6)
Haematuria (Renal and urinary disorders) | 4 (7) | 4 (5)
Renal failure (Renal and urinary disorders) | 2 (2) | 5 (5)
Urinary retention (Renal and urinary disorders) | 2 (2) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (2) | 3 (3)
Cystic haemorrhagic (Renal and urinary disorders) | 1 (1) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 21 (27)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 12 (13)
Acute respiratory failurw (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 7 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Carboxymaltose (N=1532) | Placebo (N=1533)
Pneumonia (Infections and infestations) | 57 (64) | 35 (37)
COVID-19 (Infections and infestations) | 39 (39) | 37 (39)
Sepsis (Infections and infestations) | 21 (22) | 13 (14)
Cellulitis (Infections and infestations) | 12 (12) | 21 (27)
COVID-19 pneumonia (Infections and infestations) | 11 (11) | 17 (17)
Urinary tract infection (Infections and infestations) | 17 (20) | 9 (11)
Acute kidney injury (Renal and urinary disorders) | 46 (60) | 40 (49)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 13 (14) | 15 (17)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 21 (27)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 12 (13)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 44 (54) | 45 (60)
Nervous system disorders (Nervous system disorders) | 39 (46) | 46 (55)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 43 (54) | 35 (39)
Hypotension (Vascular disorders) | 17 (17) | 15 (18)
General disorders and administration site conditions (General disorders) | 29 (34) | 31 (34)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 25 (26) | 27 (28)
Neoplasms benign, malignant and unspecified (incl systs and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (27) | 27 (31)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 15 (15)
Hepatobiliary disorders (Hepatobiliary disorders) | 17 (19) | 11 (12)
Investigations (Investigations) | 9 (11) | 17 (19)
Cardiac disorders (Cardiac disorders) | 50 (56) | 52 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT03037931/Prot_SAP_000.pdf